CLINICAL TRIAL: NCT03695978
Title: Practical Utilisation of Octapharma FVIII Concentrates in Previously Untreated & Minimally Treated Haemophilia A Patients Entering Routine Clinical Treatment With Nuwiq, Octanate or Wilate - Efficacy & Safety Observational Study-Protect-NOW
Brief Title: Efficacy, Safety & Utilisation of Nuwiq, Octanate and Wilate in Previously Untreated & Minimally Treated Haemophilia A Patients
Acronym: Protect-NOW
Status: Recruiting | Type: Observational
Sponsor: Octapharma (Industry)
Responsible Party: Sponsor
Other Study IDs: GENA-25
Record Dates: First submitted 2018-10-03; First posted 2018-10-04 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Haemophilia A
MeSH Terms: conditions — Hemophilia A

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Nuwiq: All patients receiving Nuwiq (recombinant FVIII)
- Octanate: All patients receiving Octanate (plasma derived FVIII)
- Wilate: All patients receiving Wilate (plasma derived FVIII/von Willebrand factor [VWF])

SUMMARY:
International, post-authorisation non-interventional study to evaluate real-life effectiveness, safety and utilisation patterns of Octapharma's FVIII concentrates Nuwiq, Octanate, and Wilate in previously untreated and minimally treated severe haemophilia A patients in routine clinical practice.

DETAILED DESCRIPTION:
Octapharma's FVIII concentrates have been tested in clinical trials and registered for treatment of haemophilia A; however, as haemophilia A is a rare disease, the numbers of patients treated in studies so far are limited. For previously untreated patients (PUPs), who are typically young children, and for minimally treated patients (MTPs), who have been exposed to only minimal FVIII dosages, there is a general interest to increase the body of data on treatment effectiveness and safety, particularly related to inhibitor development. Also, specifically for PUPs, treatment algorithms are not standardized, e.g. with respect to utilisation, dosage, frequency or optimal start age of FVIII prophylaxis. Real world evidence derived from a non-interventional study (NIS) can describe product utilisation and demonstrate value over a product's life cycle and facilitate benefit-risk assessments. The purpose of this study is thus to evaluate product utilisation, effectiveness and safety, including inhibitor development information, in severe haemophilia A PUPs and MTPs, who have been prescribed Octapharma's FVIII concentrates.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients of any age and ethnicity
* Severe haemophilia A (FVIII:C<1%)
* Decision to prescribe Octapharma's FVIII concentrate before enrollment into the study
* Either
* No previous treatment with FVIII concentrates or other blood products containing FVIII (PUPs) OR
* Less than 5 Exposure Days (EDs) to FVIII concentrates or other blood products containing FVIII (MTPs), if
* data are available on all previous treatment, AND
* they did not develop an inhibitor at any time point, OR
* they developed an inhibitor during treatment with an Octapharma FVIII concentrate AND continue treatment with THIS Octapharma FVIII concentrate (in the presence or absence of emicizumab).
* Voluntarily given, fully informed written and signed consent obtained before any study-related data documentation is conducted (obtained from the patient's parent/legal guardian)

Exclusion Criteria:

* Diagnosis with a coagulation disorder other than haemophilia A
* Concomitant treatment with any systemic immunosuppressive drug
* Participation in an interventional clinical trial during the time period evaluated
* Participation in another non-interventional study of Octapharma

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: A total of 200 patients, either previously untreated patients (PUPs) or minimally treated patients (MTPs), are planned to be documented in the study
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2018-02-13 (Actual); Primary Completion 2030-06 (Estimated); Study Completion 2030-06 (Estimated)

PRIMARY OUTCOMES:
Annualised rate of breakthrough bleeds to assess efficacy in prophylactic treatment | 100 exposure days
  Annualised rate of all bleeding events (BEs), including all spontaneous, traumatic and joint BEs
Incidence of Adverse Drug Reactions (ADRs) | 100 exposure days
  Adverse drug reactions (ADRs) including hypersensitivity reactions will be recorded in by patients in treatment diaries, which will be reviewed at each Follow-up Visit.

SECONDARY OUTCOMES:
Dosage of FVIII concentrates | 100 exposure days
  For each individual FVIII injection the dose will be recorded.
Overall assessment of the effectiveness of surgical prophylaxis by the treating physicians | 100 exposure days
  At the end of the postoperative period, treating physicians will assess the effectiveness of surgical prophylaxis using a scale including the four items: 'excellent,' 'good,' moderate,' and 'none'.

CONTACTS AND LOCATIONS:
Overall Officials: Sigurd Knaub, PhD, Study Director — Octapharma
Locations (54):
- United States (3):
  - University of Miami Miller School of Medicine, Miami, Florida
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Cure 4 The Kids Foundation Children's Specialty Center, Las Vegas, Nevada
- CENIDOR, Salta, Argentina
- Azerbaijan State Advanced Training Institute for Doctors Hematology Department Scientific-Research Center of Hemophilia, Baku, Azerbaijan
- Belarus (2):
  - Republican Scientific Center for Radiation Medicine and Human Ecology, Homyel
  - Republican Scientific and Practical Centre of Children Oncology, Hematology and Immunology, Minsk
- Belgium (2):
  - Hôpital Universitaire des Enfants Reine Fabiola, Brussels
  - Cliniques Universitaires Saint-Luc, Brussels
- Canada (2):
  - McMaster University, Division of Pediatric Hematology/Oncology Room 3N27, Hamilton, Ontario
  - Department of Hematology Research Research Transition Facility, Edmonton
- University Hospital Centre Zagreb, Zagreb, Croatia
- Tallinn Childrenś Hospital Clinic of Paediatric Department of Haematology and Oncology, Tallinn, Estonia
- France (7):
  - CENTRE HOSPITALIER UNIVERSITAIRE de BESANCON, Besançon
  - CHRU Tours - Hôpital Trousseau, Chambray-lès-Tours
  - Centre Régional de Traitement de l'hémophilie, Le Mans
  - Hopital Simone Veil Groupement Hospitalier Eaubonne-Montmorency, Montmorency
  - CHU Hotel Dieu, Centre de Traitment de l'Hemophilie, Nantes
  - Hôspital Necker Enfants Malades, Paris
  - CHRU Hopital Nord, Secretariat de pediatre, bat E niv +3, Saint-Priest-en-Jarez
- Germany (5):
  - Vivantes - Netzwerk für Gesundheit GmbH Klinikum im Friedrichshain, Berlin
  - Institute of Experimental Haematology and Transfusion Medicine (IHT) University Clinic Bonn (AöR), Bonn
  - Coagulation Research Centre GmbH, Duisburg
  - University Hospital Essen, Essen
  - HZRM GmbH, Frankfurt
- Hungary (2):
  - Heim Pál National Pediatric Institute Department of Oncology and Hematology, Budapest
  - University of Debrecen Department of Pediatrics, Debrecen
- Italy (11):
  - Ospedale Pediatrico "Giovani XXIII", Bari
  - Policlinico Sant'Orsola Malpighi, Bologna
  - Ospedale San Giacomo, Castelfranco Veneto
  - Azienda Ospedaliera-Universitaria Policlinico "Vittorio Emanuele", Centro di Riferimento Regionale per la Prevenzione, Diagnosi e Cura delle Malattie Rare della Coagulazione nel Bambino e neel'Adulto. U.O.C Ematologia con trapianto di Midollo Osseo, Catania
  - Azienda Ospedaliero Universitaria Careggi, Florence
  - Ospedale Maggiore Policlinico, Milan
  - Center for Thrombosis and Hemorrhagic Diseases, IRCCS Humanitas Research Hospital, Milan
  - Centro Emofilia - AUO di Padova, Padua
  - Policlinico Umberto I, Rome
  - C.tro Emofilia A.O. Città della salute e della scienza di Torino, Ospedale Regina Margherita, Torino
  - Ospedale Regina Margherita, Turin
- Children's Hospital Affiliate of Vilnius Universtity Hospital Santaros Klinikos, Vilnius, Lithuania
- Mexico (3):
  - Hospital Infantil de Morelia Eva Sámano de López Mateos, Morelia
  - Hospital Universitario Dr. José Eleuterio Gonzalez S/N, Nuevo León
  - SMO and Scientific Services S.A.P.P de C.V, Nuevo León
- Russia (2):
  - Moscow State Government-financed Public Healthcare Institution "Morozovskaya Children Clinical Hospital of Moscow Healthcare Department", Moscow
  - Saint-Petersburg State Budget Healthcare Institution "City Out-patient Clinical # 37", Saint Petersburg
- Spain (5):
  - Hospital General Universitario de Alicante Hematología y Hemoterapia, Alicante
  - Hospital Universitari Vall D'Hebrón, Unitat d'Hemofilia, Barcelona
  - HRU Malaga, Málaga
  - Universitary Hospital Son Espases (Hematology Service), Palma de Mallorca
  - Hospital Universitario y Politécnico La Fe, Valencia
- Istanbul University Faculty of Medicine, Fatih, Turkey (Türkiye)
- United Kingdom (4):
  - John Radcliffe Hospital, Oxford University Hospitals, NHS Foundation Trust, Headington, Oxford
  - Birmingham Children's Hospital NHS Foundation Trust, Birmingham
  - Great Ormond Street Hospital for Children NHS Trust, Haemophilia Centre, London
  - Newcastle Haemophilia Comprehensive Care Centre, Royal Victoria Infirmary, Newcastle upon Tyne

REFERENCES:
- [Derived] Oldenburg J, Halimeh S, Hall GW, Klamroth R, Vera PM, Jansen M, Mathias M. Design of a Real-World Observational Study in Previously Untreated and Minimally Treated Hemophilia A Patients: Protect-NOW. TH Open. 2023 May 10;7(2):e110-e116. doi: 10.1055/s-0043-1768464. eCollection 2023 Apr. PMID 37180427